CLINICAL TRIAL: NCT01570855
Title: Chemotherapy Resistance and Sensitivity Testing in Lung Tumors
Status: Completed | Type: Observational
Sponsor: Marshall University (Other)
Collaborators: Cabell Huntington Hospital (Other)
Responsible Party: Principal Investigator, Pier Paolo Claudio, M.D., Ph.D., Associate Professor of Biochemistry and Microbiology, Marshall University
Other Study IDs: 246601-1
Record Dates: First submitted 2012-03-19; First posted 2012-04-04 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Lung Cancer
Keywords: Lung cancer; chemosensitivity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to screen chemotherapy drugs currently used to treat lung cancer and determine the most effective treatment based on results of chemo sensitivity testing on the patients own cancer cells in the laboratory. The results of this screening will not influence the patients treatment.

DETAILED DESCRIPTION:
The chemosensitivity assay will be performed on tissue obtained during the diagnostic fine needle aspiration, core biopsy, or excisional biopsy of the lung lesion. Cancer cells (Bulk of tumor) and Cancer Stem Cells (CSCs) will be isolated and expanded in the laboratory.

The drug screening assay will be used to evaluate the response of the CSCs and of the cancer cells to the various chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed diagnosis of lung cancer

  * undergoing a fine needle aspiration, core biopsy, or excisional biopsy for diagnosis.
* Chemotherapy must be clinically indicated for treatment of the patient's qualifying disease
* Patient must be at least 18 years of age
* Patient must have signed an IRB approved informed consent form for the data collection study prior to entry of data into the enrollment form in the database.

Exclusion Criteria:

* Patient pathology shows benign pathology for sample submitted
* Patient is not indicated to receive chemotherapy for their disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a suspected or confirmed diagnosis of lung cancer, and who are scheduled to have a diagnostic fine needle aspiration, core needle biopsy, or excisional biopsy of the lung lesion.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tumor size | 3 months
  Tumor response will be evaluated (progression/regression) by CT scan at 3 months from therapy start.
  Clinical response to chemotherapy of lung cancer tumor cells versus lung cancer stem cells to standard of care chemo drugs will be evaluated and correlated to predicted drug by ex vivo assay.

CONTACTS AND LOCATIONS:
Overall Officials: Pier P. Claudio, M.D., Ph. D, Principal Investigator — Marshall University School of Medicine
Locations (1):
- Cabell Huntington Hospital, Huntington, West Virginia, United States